CLINICAL TRIAL: NCT03341481
Title: Effectiveness of a Dietary Supplement Femaltiker in Improvement of Initiation and Stimulation Lactation Among Mothers of Preterm Infants
Brief Title: Effectiveness of Femaltiker in Stimulation Lactation Among Mothers of Preterm Infants
Acronym: FEMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Human Milk Bank Foundation (Unknown); Nutropharma LLC (Unknown)
Responsible Party: Principal Investigator, Maria Katarzyna Kornacka, Professor of Neonatology, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FEMA/01/2014
Record Dates: First submitted 2017-03-23; First posted 2017-11-14 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2017-11

CONDITIONS: Lactation Induced
Keywords: galactagogues, lactogenesis, preterm labor
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Intervention Model Description: Treatment was given to the mothers assigned to the galactogogue group, whereas a placebo was given to those assigned to the placebo group. Each patient randomized to either treatment or placebo group received 28 sachets for 14 days of the trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: To mask intervention the placebo was used. In this case, the placebo was prepared as a blend of sucrose, apple fiber and natural aroma caramel by subcontractor of the producer, accordingly to the GMP (number of sachets prepared 1534). Placebo sachets were in the same size sachets as the product and could be hardly distinguished in term of color, taste or texture and flavor. To the end of the trial patients and medical staff were blinded which sachet contained active product. People responsible for the data clean-up and statistics were partially blinded since theyhad to know which patients were in the same treatment group.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Femaltiker (Experimental): 7.7 g of Femaltiker twice a day for 14 days of the trial.
  Interventions: Other: Femaltiker
- placebo (Placebo Comparator): 7.7 g placebo 14 days of the trial.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Femaltiker — Patient had taken twice a day the product
  Other Names: LACTANELL formula
  Arms: Femaltiker
Other: Placebo — Patient had taken twice a day the placebo
  Arms: placebo

SUMMARY:
Femaltiker is a food for special medical purposes with a unique composition. Because beer, but not ethanol, has been reported in a number of studies to stimulate prolactin levels and breastmilk production, polysaccharide from barley was chosen as a potential galactogogue. To verify our assumption, a randomized, double blinded research with placebo was performed. The study was conducted according to good clinical practice and 10% of output data was audited by the outside monitor. The research was conducted from 14 April 2014 to 7 October 2015 in two NICUs with consent of the ethics committee on Medical Warsaw University.

DETAILED DESCRIPTION:
The traget population consisted of volunteers women who delivered infants at < 37 weeks gestation. Criteria of exclusion were: hypothyroidism and diabetes type I or II diagnosed and treated before pregnancy.

The schedule of the study included three visits with in certain point time during two weeks postpartum. During the study patients had taken twice a day product or placebo, respectively. The protocol of the study included :

* Three consecutive blood collections for examination of prolactin level on every visit (10 min beforeBlood examination of prolactin level in triplet on every visit (10 min before breastfeeding session, 10 min after beginning of breastfeeding and 10 min. after finishing of breastfeeding.)
* Filling pumping log to control variation in the milk yield and efficacy of lactation.
* Measurement of the volume of milk producing before blood examination (directly in case of pumping by the mother or indirectly based on weight of the baby before and after feeding)
* Interview with lactation consultant concerning patient's self-estimation of lactation efficacy Data collection was done using the CRF in the paper form which were then put tto the database in ExcelDocuments.

ELIGIBILITY:
Inclusion Criteria:

* mothers of preterm infants (born before 37 completed weeks of pregnancy)

Exclusion Criteria:

* hypothyroidism
* diabetes type I or II diagnosed and treated before pregnancy
* participating in other study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2014-04; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
The volume of milk produced by study participants | two weeks after delivery
  Measurement of the volume of expressed milk
Level of serum prolactin | two weeks after delivery
  Three consecutive blood collections for prolactin level

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Wesolowska, PhD, Study Director — Warsaw Medical University, Department of Neonatology; Maria K. Borszewska-Kornacka, Prof., Principal Investigator — Warsaw Medical University Hospital, Department of Neonatology and Intensive Care Unit
Locations (4):
- Poland (4):
  - Warsaw Medical University Hospital, Warsaw
  - Mother and Child Health Center of Warsaw Medical University, Warsaw
  - Laboratory of Human Milk and Lactation Research at Regional Human Milk Bank in Holy Family Hospital, Warsaw
  - Warsaw Medical University - Clinic of Neonatology, Warsaw

IPD SHARING:
Plan to Share IPD: No